CLINICAL TRIAL: NCT03086720
Title: Effect of Sodium Hypochlorite Pre-treatment on the Retention of Restorations for Non-carious Cervical Lesions: A Randomized Controlled Trial
Brief Title: Deproteinization as a Coadjuvant in Dentin Adhesion of Noncarious Cervical Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPEL- PPGO 0019
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Non-carious Cervical Lesions
Keywords: Adhesive system; Controlled clinical trial; Dental restoration; Noncarious cervical lesions; Dental restoration failure; Sodium hypochlorite
MeSH Terms: interventions — Sodium Hypochlorite; Water

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium hypochlorite (Experimental): Dentin pre-treatment with a experimental solution (sodium hupochlorite), after the dentin acid etching
  Interventions: Procedure: Sodium hypochlorite
- Water (Placebo Comparator): Application of water (placebo) after dentin acid etching
  Interventions: Procedure: Water

INTERVENTIONS:
Procedure: Sodium hypochlorite — Application of 10% sodium hypochlorite (60 seconds) after the etching procedure and before the adhesive system.
  Arms: Sodium hypochlorite
Procedure: Water — Treatment of acid etched dentin with sterilized water for 60 s before adhesive system application
  Arms: Water

SUMMARY:
This study will verify the effect of the application of a substance (10% sodium hypoclorite -NaOCL) in dentin on noncarious cervical lesions, with the aim of increasing the longevity of the restorations performed in this type of lesion.

The hypothesis of the present study is that the application of deproteinization solution after acid etching does not influence the failure rate of the restorations.

DETAILED DESCRIPTION:
The purpose of this study will be to evaluate the failure rates of composite restorations of non-carious cervical lesions (NCCL) performed with or without the pre-treatment with 10% sodium hypochlorite (NaOCl) on etched dentin.

A randomized controlled split-mouth and double blind clinical trial will be carried out. Patients with at least two NCCL will be selected. Each patient will be received at least one pair of composite restorations (Filtek Z350/3M ESPE), bonded either with 2 techniques: control (acid etching + placebo solution for 60 seconds + Adper Single Bond 2/3M ESPE) or experimental (acid etching + 10% NaOCl for 60 seconds + Adper Single Bond 2). A calibrated examiner will be evaluated the restorations (baseline, 6-, 12-, 24- and 36-month) using the FDI criteria. The primary outcome is retention of the restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at least two non-carious cervical lesions (NCL) in anterior, canine or pre-molars;
* Patients who had more than 20 teeth in the mouth;
* Patients who were at least 18 years of age at the time of treatment and capable to understand and sign the written informed consent;
* NCL in the facial surface of the teeth with sometimes a small part extending interproximally; Patients with good periodontal heath.

Exclusion Criteria:

* Patients with smoking habits, practicing bruxism, severe systemic diseases, using active orthodontic treatment, malocclusion (Angle Class II or Class III);
* Tooth with the NCL with the absent of antagonist;
* NCL wear facets upper than 50% of the incisal/occlusion surface, as a result of tooth attrition;
* Presence of caries or restorations in the area to be treated;
* Full-mouth visible plaque index (VPI) or full-mouth gingival bleeding index upper than 20%, probing depth and clinical attachment loss values exceeding 4 mm with bleeding on probing;
* Unwillingness to return for follow-ups or refuse to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Retention rates of the restoration | 6, 12, 24, 36 and 60 months
  Patients will be reevaluated at each specified time point and all restoration sites will be evaluated to check if the restoration will be still in place, or if it is missing, or if there is partial retention

SECONDARY OUTCOMES:
Change from baseline in Post-operative sensitivity | 6, 12, 24, 36 and 60 months
  At each time-point, patients will be recalled and interviewed regarding any symptom related to each restorations placed.
Change from baseline in marginal staining rates | 6, 12, 24, 36 and 60 months
  At each time-point, patients will be recalled and restorations will be reassessed in order to record changes in the rates of marginal staining, using the World Dental Federation (FDI) criteria for restorations assessment (Hickel et al 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano Cenci, PhD, Principal Investigator — School of Dentistry, Federal University of Pelotas
Locations (1):
- Federal University of Pelotas - School of Dentistry, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Favetti M, Schroeder T, Montagner AF, Correa MB, Pereira-Cenci T, Cenci MS. Effectiveness of pre-treatment with chlorhexidine in restoration retention: A 36-month follow-up randomized clinical trial. J Dent. 2017 May;60:44-49. doi: 10.1016/j.jdent.2017.02.014. Epub 2017 Feb 22. PMID 28237629
- [Derived] Favetti M, Schroeder T, Montagner AF, Moraes RR, Pereira-Cenci T, Cenci MS. NaOCl Application after Acid Etching and Retention of Cervical Restorations: A 3-Year Randomized Clinical Trial. Oper Dent. 2022 May 1;47(3):268-278. doi: 10.2341/20-166-C. PMID 35584331